CLINICAL TRIAL: NCT04619485
Title: Sexual and Vaginal Health in Breast Cancer Women Receiving Aromatase Inhibitors Before and After CO2 Laser Therapy: A Randomized, Double-blind, Sham-controlled Trial - LIGHT Study
Brief Title: Sexual and Vaginal Health in Breast Cancer Women Receiving Aromatase Inhibitors Before and After CO2 Laser Therapy
Acronym: LIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Inmaculada Alonso, MD, PhD, Principal Investigator, Clinical Professor, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCB/2019/0786
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Genitourinary Syndrome of Menopause
Keywords: BREAST CANCER; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Breast Neoplasms | interventions — Lasers, Gas

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAM LASER (Sham Comparator): Group A: Arm using basal treatment and adding vaginal laser using double blind to adjust the treatment to zero potence.
  Interventions: Device: CO2 SHAM LASER
- EFFECTIVE LASER (Active Comparator): Group B: Arm using basal treatment and adding vaginal laser using double blind to adjust the treatment to regular potence.
  Interventions: Device: CO2 LASER

INTERVENTIONS:
Device: CO2 LASER — 5 SESSIONS OF CO2 VAGINAL LASER
  Arms: EFFECTIVE LASER
Device: CO2 SHAM LASER — 5 SESSIONS OF CO2 VAGINAL SHAM LASER
  Arms: SHAM LASER

SUMMARY:
Background: Vulvovaginal health, directly linked to sexual health, is a key factor for female pleasure. BCS receiving AI are likely to present severe GSM and sexual complaints. Innovative options, as vaginal laser therapy, are emerging to treat GSM and sexual dysfunctions. Nowadays, data in BCS is scarce, moreover, few studies included patients receiving AI [16]. Different meta-analysis [17-23] found GSM [24, 25] and sexual function [9, 10] may improve significantly at short-term, however, the body of evidence is of low quality. Therefore, before recommendation of laser therapy for sexual complaints in BCS with GSM, there are unmet needs to be solved: efficacy and safety at long-term, biases related to patients' expectations and a detailed assessment of the complex underpinnings of sexuality.

Aims: To evaluate sexual and vaginal health in BCS receiving AI with GSM, before and after CO2 laser therapy compared to a sham-controlled group.

Methods: Prospective, randomized, double-blind controlled study with two parallel study arms: 1) Fractional CO2 laser therapy (5monthly sessions). 2) Sham laser therapy (5monthly sessions). After end-treatment, patients are followed up at 1 month and 6 months. BCS treated or undergoing AI with GSM and sexual function impairment, will be suitable. All patients will maintain first-line non-hormonal treatment and sexual assessment (PLISSIT Model) according with usual care. The primary outcome is improvement in sexual function (FSFI total score). As secondary outcomes: resumption sexual activity, sexual activity frequency, dyspareunia (VAS), female sexual dysfunction, sexual dimensions (FSFI), body image (S-BIS), quality of life (SF-12), vaginal pH acidification, maturation index and Vaginal Health Index of Gloria Backmann, adverse events, satisfaction (Likert scale) and adherence to treatment.

Expected impact: Emergent, non-invasive, laser therapy has significant benefit for BCS with AI, improving subjective and objective sexual and vaginal health outcomes and adding value to the usual care multidisciplinary approach.

DETAILED DESCRIPTION:
BACKGROUND:

Sexuality is a central aspect of being human throughout life encompasses sex, gender identities and roles, sexual orientation, eroticism, pleasure, intimacy and reproduction. Most of these aspects may be affected in breast cancer survivors (BCS). In a recent meta-analysis, focused on sexual function through Female Sexual Function Index (FSFI) among BCS, female sexual dysfunction prevalence was 73,4% (95 % CI 64-82.8 %, I2 = 96.8 %) and mean FSFI 19.28 (95 % CI 17.39-21.16, I2 = 97.6 %). Several modifiable risk factors for sexual dysfunction in BCS may be optimum targets for intervention: amelioration of vaginal discomfort and urinary incontinence, the benefits of breast conserving surgery on body image or the evaluation of relationship quality. Due to the multifaceted nature of the factors affecting sexuality in BCS, most authors encouraged the need for comprehensive assessment and for a multidisciplinary approach.

BC diagnosis and/or its treatments (surgery, chemoradiotherapy, hormonal therapy) may altered sexual health. Vulvovaginal health, directly linked to sexual health, is a key factor for female pleasure. Genitourinary syndrome of menopause (GSM) is caused by decline in estrogen at menopause, which may also appear or worsen after systemic cancer treatments as aromatase inhibitors (AI). GSM is associated with sexual symptoms (lack of lubrication, discomfort or pain, impaired function), genital symptoms (dryness, burning, irritation) and urinary symptoms (urgency, dysuria, recurrent urinary tract infections). BCS receiving AI are one of the groups most likely to present severe GSM and sexual complaints. A cross-sectional study on 129 BCS during the first 2 years of adjuvant AI therapy, found 3 out of 4 women were distressed about their sexual problems. Only 52% of women had been sexually active when endocrine therapy began, but 79% of that group developed new sexual problems.

The first line of treatment for GSM is non-hormonal therapy (regular sexual activity, moisturizers-lubricants, pelvic-floor relaxation techniques, dilators) although in many women these options will not adequately control symptoms. Hormonal therapies must be used with caution in women with estrogen-dependent cancers. So, alternative options are emerging for this subset of patients, such as vaginal laser therapy. Different studies provided short-term data on non-cancer patients that showed laser therapy was feasible, safe and improved objective and subjective GSM. Data regarding sexuality derived from secondary endpoints and suggested that laser therapy may improve sexual function, mainly decreasing sexual pain. To date, data on laser therapy in BCS is scarce, moreover, few studies included patients receiving ongoing AI. The CO2 laser was the most frequently used device. Different reviews and meta-analysis found GSM and sexual function may improve significantly at short-term, however, the body of evidence is of low quality. Therefore, before recommendation for the use of laser therapy for sexual complaints in BCS with GSM, there are unmet needs to be solved as efficacy and safety at long-term, biases related to patients' expectations of therapy and a detailed assessment of the complex underpinnings of sexuality.

AIMS:

To answer the unmet needs previously mentioned, the aim of the current study is to verify the outcomes of sexual and vaginal health in breast cancer women receiving AI, who were experiencing symptoms of GSM, before and after CO2 laser therapy compared to a sham-controlled group.

Specifically, we will compare the following subjective and objective measurements of sexual and vaginal health:

MAIN GOAL: Report an improvement in sexuality:

* Primary outcome: sexual function (FSFI total score)
* Secondary sexual outcomes: resumption sexual activity (sexually active vs non-sexually active), sexual activity frequency (nº sexual activity/week), dyspareunia (VAS), female sexual dysfunction (VAS sexual life distress), sexual dimensions: desire, arousal, lubrication, orgasm, satisfaction and pain (FSFI) and body image (S-BIS)

OTHER OBJECTIVES: Report an improvement on GSM symptoms (efficacy) and quality of life, feasibility and safety of laser therapy in BCS:

- Secondary non-sexual outcomes: quality of life (SF-12). Verify an acidification of the vaginal pH, an improvement in the maturation index and an improvement in the Gloria Backmann Index: Vaginal Health Index. To evaluate toxicity associated with vaginal laser therapy in this population (AEs and SAEs). To determine how many women with the defined patient eligibility will complete all treatments.

METHODS:

DESIGN: Prospective, randomized, double-blind controlled study with two parallel study arms: ARM I: Patients undergo fractional CO2 laser therapy at 5 times points 30 days apart. ARM II: Patients undergo sham laser therapy at 5 time points 30 days apart. After completion of the treatment, patients are followed up at 1 month and 6 months.

RANDOMIZATION PROCESS: A randomization list will be generated in multiple blocks of 2 and 1: 1 ratio with STATA version 15.1 or higher.

STUDY SUBJECTS: Patients treated or undergoing AI for BC in the Breast Cancer Unit of the Hospital Clínic and who present symptoms related to GSM that condition their sexual function and quality of life, despite receiving first-line non-hormonal treatment: regular sexual activity (such as mutual and self-touch masturbation, manual or vibrator stimulation, oral sex, sexual intercourse, massage and other forms of physical intimacy), moisturizers, lubricants, pelvic-floor relaxation techniques and/or dilators. Inclusion and exclusion criteria are summarized in Table 1.

STUDY GROUPS: All patients will receive instructions to maintain first-line non-hormonal treatment, as well as sexual assessment using the PLISSIT Model according with usual care in our hospital.

The study group will be treated with a vaginal fractionated CO2 laser protocol (The SMARTXIDE TOUCH (Deka) equipment with an autoclavable vaginal probe following the manufacturer's protocol.

The control group will receive treatment with a sham-CO2 laser using a double-blinded protocol.

STUDY STRUCTURE.

SAMPLE CALCULATION Considering FSFI score as the main variable of the study, a sample size of 22 subjects for each group was calculated, accepting an alpha risk=0.05 and a beta risk <0.1 in a bilateral contrast. The common standard deviation was considered to be of 8 points and the minimum expected effect size of 6 points. Considering follow-up loss rate of 15%, the sample size should be 51 patients.

STATISTIC ANALYSIS Descriptive statistics will be used according to standard calculation methods. The comparison between the two treatments at the end of the study will be evaluated through the change with the baseline using a mixed repeated measures model (MMRM) adjusted for the baseline value and including the treatment and the time in the model.

The variables of repetitive evaluation over time are analyzed according to the following strategy: (a) continuous variables with a repeated measures mixed longitudinal model (MMRM); (b) binary or non-normal variables with marginal models (Generalized Estimating Equation: GEE). Other variables will be studied as follows: Fisher's exact test for categorical variables, Student's t test for continuous variables between 2 groups. Non-parametric methods for independent data (Mann-Whitney U for 2 groups or Kruskall-Wallis test for more than 2 groups) will be used if necessary. The level of statistical significance will be 5% bilateral. The main analysis will be by Intention to Treat (ITT).

IMPACT:

What would be the impact of the project on sexual medicine field when it is successfully completed? Please explain how your project fits to the specific call

The BCS receiving AI are at higher risk of developing GSM symptoms. Sexual issues are common, either secondary to painful sex or as a direct effect of estrogen deprivation in the brain. However, addressing sexual health issues in BCS still meets several barriers from both, patient and health care professionals. GSM symptoms do not put survival at risk, however, have a significant impact in the quality of life.

The first-line treatment for GSM symptoms should be non-hormonal therapies according clinical guidelines, although frequently it will be insufficient to alleviate symptoms. Hormonal therapies are not currently recommended and must be used with caution in BCS. So, energy-based treatments have emerged as a promising option in this subgroup of patients. However, the body of evidence is lacking to make decisive recommendations [18], specially to treat sexual complaints. There is an urgent need to carry out RCT with larger sample size, long-term follow-up and blinded control group for answer various unmet needs in this field: short/mid and long-term safety issues and efficacy, treatment modalities (type of laser) and protocols (laser parameters, sessions numbers, repetitions).

This project aims to demonstrate that emergent, non-invasive, non-anesthetic laser therapy has significant benefit for BCS with AI, measured in a prospective, randomized, double-blind controlled trial using validated tools for subjective and objective sexual and vaginal health outcomes and quality of life.

Moreover, sexual health is a state of physical, emotional, mental and social well-being in relation to sexuality which requires the possibility of having pleasurable and safe sexual experiences. So, both arms of study groups will benefit from multidisciplinary approach including non-hormonal therapies (regular sexual activity, moisturizers, lubricants, pelvic floor relaxation techniques and/or dilators) and sexual assessment using the PLISSIT Model according with usual care in our hospital and with international recommendations.

ELIGIBILITY:
Inclusion Criteria:

* BC treated with aromatase inhibitors ± GnRH analogues (aGnRH)
* Menopause (natural or induced) and signs / symptoms of GSM
* Vaginal pH ≥5
* Negative Human Papillomavirus (HPV) cytology and / or determination
* Intention or willingness to have sex
* Signed informed consent

Exclusion Criteria:

* Vaginal hormonal treatment in the last 6 months
* Vaginal moisturizers and / or lubricants during the 30 days prior to study treatment
* Laser treatment, radiofrequency, hyaluronic acid, lipofilling in the vagina during the last 2 years
* Ospemifene treatment
* Being affected for: active infection of the genital tract; intraepithelial neoplasm of cervix, vagina, or vulva; have or have been treated for genital cancer
* Genital prolapse stage ≥II.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 12 months
  The 19 items of the FSFI use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning on the respective item. To score the measure, the sum of each domain score is first multiplied by a domain factor ratio (0.6 for desire; 0.3 for arousal; 0.3 for lubrication; 0.4 for orgasm; 0.4 for satisfaction; and 0.4 for pain) in order to place all domain totals on a more comparable scale, and then subsequently summed to derive a total FSFI score.

SECONDARY OUTCOMES:
Vaginal pH | 12 months
  Level of vaginal fluid pH
Vaginal epithelium thickness | 12 months
  Measured by Vaginal ultrasound/vaginal biopsy.
Resumption of sexual activity | 12 months
  Sexually active vs non-sexually active
Sexual activity frequency | 12 months
  Number of sexual activity /week
Dyspareunia | 12 months
  Measured by Visual Analogue Scale
Female sexual dysfunction | 12 months
  Visual Analogue Scale of sexual life distress
Body image perception | 12 months
  Measured by S-BIS scale

CONTACTS AND LOCATIONS:
Overall Officials: Immaculada Alonso Vargas, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Eduard Mension Coll, Barcelona, Spain

REFERENCES:
- [Derived] Mension E, Alonso I, Angles-Acedo S, Ros C, Otero J, Villarino A, Farre R, Saco A, Vega N, Castrejon N, Ordi J, Rakislova N, Tortajada M, Matas I, Gomez S, Ribera L, Castelo-Branco C. Effect of Fractional Carbon Dioxide vs Sham Laser on Sexual Function in Survivors of Breast Cancer Receiving Aromatase Inhibitors for Genitourinary Syndrome of Menopause: The LIGHT Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255697. doi: 10.1001/jamanetworkopen.2022.55697. PMID 36763359

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04619485/Prot_SAP_001.pdf